CLINICAL TRIAL: NCT05039099
Title: A Phase 2a, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate Safety, Tolerability, Pharmacodynamic Markers, and Pharmacokinetics of AP-101 in Patients With Familial Amyotrophic Lateral Sclerosis (fALS) and Sporadic Amyotrophic Lateral Sclerosis (sALS)
Brief Title: A Study to Evaluate, Safety, Tolerability, Pharmacodynamic (PD) Markers and Pharmacokinetics (PK) of AP-101 in Participants With Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AL-S Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP101-02; 2020-005971-11 (EudraCT Number)
Record Dates: First submitted 2021-09-01; First posted 2021-09-09 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Familial Amyotrophic Lateral Sclerosis; Sporadic Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Amyotrophic lateral sclerosis 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AP-101 (Experimental): AP-101 is administered by IV.
  Interventions: Drug: AP-101
- Placebo (Placebo Comparator): Placebo is administered by IV.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AP-101 — Participants receive AP-101 by intravenous infusion (IV).
  Arms: AP-101
Drug: Placebo — Participants receive placebo by IV.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, PK, and PD of AP-101 in participants with fALS and sALS.

ELIGIBILITY:
Inclusion Criteria:

* All participants must adhere to contraception restrictions
* Female participants of childbearing potential must adhere to contraception restrictions
* Have possible, clinically probable, clinically probable-laboratory supported or definite familial or sporadic ALS in accordance with the El-Escorial criteria or who have a diagnosis of ALS as defined by the Gold Coast Criteria; progressive motor impairment documented by history or repeated clinical examination, preceded by normal motor development, and presence of upper and lower motor neuron dysfunction in at least 1 body region or lower motor neuron dysfunction in at least 2 body regions and investigations excluding other conditions
* In familial ALS participants, a confirmed pathogenic superoxide dismutase 1 (SOD1) mutation
* Onset of symptoms (i.e, weakness) within past 24 months prior to screening, at the time of obtaining informed consent
* Have slow vital capacity (SVC) of greater than or equal to (> or =) 50 percentage (%) of predicted values. Participants with SVC of <50% of predicted values may be permitted to enter the open-label extension, based on the opinion of the investigator
* Absence of bilevel positive airway pressure (BiPAP)/proportional assist ventilation (PAV) > 4 hours for symptoms attributable to ALS. Use of a CPAP for pre-existing conditions will be allowed
* If on riluzole, must be on a stable dose.
* If on edaravone, must have completed 2 cycles and are expected to remain on the same dose throughout the study
* Able to provide informed consent which includes compliance with the requirements and restrictions
* Have venous access sufficient to allow for blood sampling
* Have clinical laboratory test results within the normal reference range for the population or study site, or results with acceptable deviations that are judged to be not clinically significant by the investigator

Exclusion Criteria:

* Have participated or currently participating in another clinical trial within 12 weeks of baseline (Day 1)
* Have undergone a tracheostomy for ALS symptoms
* Are on nasal intermittent positive pressure ventilation (NIPPV) >4 hours per day for the treatment of ALS related symptoms
* Have other causes of neuromuscular weakness
* Have cognitive impairment, severe disease in the cardiovascular, hematological, renal system, neurodegenerative disease, pulmonary disorder, or psychiatric illness
* Pregnant or nursing women
* Have been exposed to any antisense treatment targeting SOD1 within 6 months of the baseline visit
* Have undergone stem cell therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious AEs (SAEs) | From start of the study up to Week 51
  An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with the study intervention. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, other situations.
Number of Participants with Abnormalities in Vital Signs, Clinical Laboratory Assessments, Physical and Neurological Examinations, Electrocardiograms (ECGs) | From start of the study up to Week 51

SECONDARY OUTCOMES:
Elimination half-life (t1/2) of AP-101 in Serum | Predose up to Week 51
Area Under the Drug Concentration-Time Curve (AUC) | Predose up to Week 51
Concentration at End of Infusion (Cat EOI) | Week 24
Change From Baseline in AP-101 Levels in the Cerebrospinal Fluid (CSF) up to Week 24 | Baseline, up to Week 24
Change From Baseline in Neurofilament Light Chain and Phospho-Neurofilament Heavy Chain Levels in the Cerebrospinal Fluid (CSF) up to Week 51 | Baseline, up to Week 51
Change From Baseline in Neurofilament Light Chain and Phospho-Neurofilament Heavy Chain Levels in Plasma up to Week 51 | Baseline, up to Week 51

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — AL-S Pharma SA
Locations (13):
- UC San Diego, ACTRI, La Jolla, California, United States
- Department of Neurology, University Hospitals, Leuven, Belgium
- Canada (4):
  - ALS clinic at the Kaye Edmonton Clinic, University of Alberta, Edmonton, Alberta
  - London Health Sciences Centre - Victoria Hospital, London, Ontario
  - ALS Research Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Montreal Neurological Institute and Hospital / Dr Genge, Montreal, Quebec
- Germany (4):
  - Hannover Medical School, Hanover, Hanover
  - Charité, Berlin, State of Berlin
  - Ulm University Hospital, Ulm, Ulm
  - Deutsches Zentrum für Neurodegenerative Erkrankungen e.V. (DZNE), Bonn
- Hanyang University Medical Center, Seoul, Seoul, South Korea
- Sweden (2):
  - Studieenheten Akademiskt specialistcentrum, SLSO, Stockholm, Stockholm County
  - Norrlands universitetssjukhus/ University Hospital of Northern Sweden (NUS), Umeå